CLINICAL TRIAL: NCT02821767
Title: Studies of the Natural History, Pathogenesis and Outcome of Ocular Disorders
Brief Title: Natural History, Pathogenesis, and Outcome of Ocular Disorders
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160134; 16-EI-0134
Record Dates: First submitted 2016-06-29; First posted 2016-07-04 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12-19

CONDITIONS: Eye Disease
Keywords: Eye Disease; Natural History
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: subjects with diagnosed or undiagnosed ocular conditions and/or their first-degree relatives

SUMMARY:
Background:

The National Eye Institute (NEI) wants to evaluate and provide standard treatment to people with eye diseases.

Objective:

To examine and treat people with eye diseases and learn more about eye diseases and how they are inherited.

Eligibility:

People with eye diseases who can give consent or have a guardian who can consent for them. Asymptomatic first-degree relatives willing to provide a blood sample may also be enrolled for the purpose of genetic testing.

Design:

Participants will be screened with an eye exam.

Participants will have 1-12 visits per year depending on their eye disease for up to 5 years. Visits last about 4 hours and could include:

Medical and family history

Physical exam

Eye exam and photography.

Oculography: They put on contact lenses or goggles. They watch spots on a computer

screen for 20-30 minutes.

Electrooculography: Small metal disks are placed on the skin next to both eyes. They look left

and right in the dark and light for about 30 minutes.

Electroretinography: They sit in the dark with their eyes patched. A small metal disk is taped

to the forehead. After 30 minutes, the patches are removed and contact lenses put in. They

watch flashing lights.

Fluorescein angiography: A needle guides a thin plastic tube into an arm vein. A dye is

injected through the tube and travels up the blood vessels in the eyes. Pictures are taken of the

eyes.

Immunosuppressive treatment

Eye cell sample: Samples are obtained from swabbing, pressing paper on, or taking a small

biopsy sample from the surface of the eye.

Blood tests

Skin, tear, urine, saliva, stool, or hair sample

Exam under anesthesia for some children

At each visit participants could get medications, eye drops, eye injections, laser treatments, or surgery.

DETAILED DESCRIPTION:
The National Eye Institute (NEI) is conducting a study to evaluate and provide standard treatment to participants with various diagnosed and undiagnosed ocular conditions.

Objective: The primary objective of this protocol is to collect data and specimens generated

through clinical care procedures. Through this primary objective, the secondary objectives (establish a resource of patients with ocular conditions to facilitate recruitment into new research protocols at the NEI, gain additional knowledge about the course of specific ocular diseases and characterize the natural history of such diseases (to generate hypotheses for future clinical research studies), and evaluate the effects of standard of care treatments) may be achieved.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Have a diagnosed, undiagnosed or suspected eye disease.
2. Have the ability to understand and sign an informed consent or have a parent/legal guardian do so if they are minor children or a legally authorized representative to provide consent for adults without consent capacity.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Are unwilling to give informed consent or assent when applicable.
2. Are unwilling or unable to be followed as clinically indicated.
3. Have a systemic disease that compromises the ability of NEI clinicians to provide adequate ophthalmologic examination or treatment.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-08-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
No formal outcomes will be measured; however, the clinical assessments of enrolled participants can be used to measure the response to standard treatment. | ongoing
  response to standard care of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Awilda V Holland, R.N., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-EI-0134.html